CLINICAL TRIAL: NCT02439827
Title: The "Fortaleça Sua Saúde" Program: A Cluster-randomized Controlled Trial to Promote Active and Healthy Lifestyle Among Brazilian Students
Brief Title: The "Fortaleça Sua Saúde" Program for Active and Healthy Lifestyle Among Brazilian Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Catarina (Other)
Collaborators: Universidade Federal do Ceara (Other); Secretaria Municipal de Educação de Fortaleza, Ceará, Brazil (Unknown)
Responsible Party: Principal Investigator, Valter Cordeiro Barbosa Filho, Master of Science in Physical Education, PhD Student in Physical Education, Universidade Federal de Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UniversidadeFSC
Record Dates: First submitted 2015-05-03; First posted 2015-05-12 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Adolescent Behavior
Keywords: Lifestyle; Intervention; Motor Activity; Mediating Variables; Mental Health; Obesity; Adolescent Health; School; Health Promotion; Brazil
MeSH Terms: conditions — Adolescent Behavior; Motor Activity; Psychological Well-Being; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- "Fortaleça sua Saúde" program (Experimental): The intervention program was structured into four main components: (i) training and activities in general curriculum; (ii) training and activities in Physical Education classes; (iii) active opportunities in the school environment; (iv) health education in school community.
  Interventions: Behavioral: "Fortaleça sua Saúde" program
- Control (No Intervention): Schools from the control group carried out one semester with the regular and conventional activities of a full-time school. In general, the control schools had two weekly Physical Education classes that include content and activities according to the perspective of their teachers. The conventional Programa Saúde na Escola were also performed in these schools.

INTERVENTIONS:
Behavioral: "Fortaleça sua Saúde" program — The program duration was of one academic semester (approximately four months) in 2014. The intervention strategies focus on teachers' training and activities on health in curriculum (including a specific training to Physical Education teachers), active opportunities in the school environment (availability of spaces and materials for PA) and health education (production and exhibition of health material at school, and distributing pamphlets to students and parents).
  Arms: "Fortaleça sua Saúde" program

SUMMARY:
Background:

Interventions on lifestyle among adolescents are important, but the main mechanisms that explain the changes (mediating variables) on lifestyle have been little explored. Investigators present the rationale and methods of a cluster-randomized controlled trial aimed to promote promotion active and healthy lifestyle (especially physical activity [PA] practice and reducing screen time use) among Brazilian students - the "Fortaleça sua Saúde" ("Strengthen Your Health" in Portuguese) program.

Methods/Design:

This is a school-based cluster-randomized controlled trial that included students from six elementary full-time public schools (7-9 grades) in Fortaleza, northeastern Brazil. The intervention duration was one academic semester (approximately four months) in 2014. The intervention strategies focused on teachers' training and activities on health in curriculum (including a specific training to Physical Education teachers), active opportunities in the school environment (availability of spaces and materials for PA) and health education (production and exhibition of health material at school, and distributing pamphlets to patients). Data collection will be performed before and immediately after 4 months of intervention. The primary variables include the practice of PA (weekly PA volume) and the screen time use (TV/computer/video games). Intrapersonal, interpersonal and environmental variables associated to PA and screen time use will be evaluated by standardized questionnaire. Other components of the lifestyle (e.g., eating habits), psychological (e.g., self-rated health, body satisfaction), biological (general and abdominal obesity) and academic performance will be also evaluated in the patients. Depressive symptoms, eating disorders, sleep quality, objectively-measured physical activity will be evaluated in obese patients.

Discussion:

Is effective, this program will contribute to the development of public policies for active and health lifestyle promotion among young population, especially from low- and middle-income countries. The main variables (intrapersonal, interpersonal and/or environmental stimulus) that help the young people to adopt an active lifestyle also may be indicated. Finally, investigators expect that the proposed strategies may be adaptable to the public school reality and they may be extended to the entire school system.

DETAILED DESCRIPTION:
Setting and Population:

Fortaleza is the capital of Ceara state, northeastern Brazil, and has a population of 2,452,185 inhabitants (the fifth largest city in Brazil considering the population). This municipality has an area of 314 km² and a Human Development Index (HDI) of 0.754. The city of Fortaleza is geographically divided into six administrative regions.

According to the Municipal Education Department, forty schools attended 6-9 grades and included the Programa Saúde na Escola, and six out of these schools had a full-time education model. These six schools attended approximately 2,500 students, of which 1,272 were enrolled in classes from 7th to 9th grades.

These six schools had similar characteristics (e.g., size, target audience, curriculum, etc.) and were located in different administrative regions (geographically disperses). Therefore, there was no need to conduct peer schools during random selection to prevent study contamination. Three schools were randomly selected to intervention group and other schools were control group. The neighborhood-HDI from where the six schools were located was similar between groups (neighborhood-HDI of 0.215, 0.341 and 0.443 for intervention schools, and 0.170, 0.377 and 0.491 for control schools).

Theoretical basis of the "Fortaleça sua Saúde" program:

The "Fortaleça sua Saúde" program was structured considering different theoretical aspects. The Socioecological Theory emphasizes that intrapersonal (e.g., knowledge, self-efficacy), interpersonal (social support, peer and family model) and environmental (perception and environmental characteristics) aspects interfere independently and interactively in the individual's behavior. The actions of the program "Fortaleça sua Saúde" program were directed to achieve these different levels. The concepts of the Health Promoting in Schools was also used. Three characteristics were used in order to choice the program components: Health education topics in the formal school curriculum, health values, attitudes and opportunities promoted within the school, and schools seek to engage with families, outside agencies and the wider community.

Description of the Intervention:

The "Fortaleça sua Saúde" intervention during the second scholar semester (approximately four months).

Training and activities in general curriculum:

All teachers from three intervention schools were invited to participate of training and to execute class activities focused on the discussion of active and healthy lifestyle. Full training was structured in three stages (two face-stages and one distance-stage) with certification recognized by the University.

A four-hour training were performed at the beginning of school semester. Discussions on primary health concepts and the importance of these issues were made, including the relationship between health, school and academic performance. Proposals for cross-cutting issues including the National Curriculum Standards were also discussed. Finally, strategies directed to combine teaching tools (e.g., homework, tests presentations) and health issues (e.g., physical activity [PA], quality of life, health eating) were discussed.

Teachers received a supplemental manual in order to help the classroom activities. This manual was prepared by program staff based on other productions on health in school, but they were adapted to the reality of Fortaleza's schools and students. Brazilian documents on education were consulted including the Learning Expectations of the Municipal Education Department and the National Curriculum Standards on health topics. Ministerial reports on health and education were also consulted. The manual included proposals for activities according to knowledge areas (i.e., languages, social sciences, natural sciences and mathematics). For example, in mathematics, an included proposal was about teaching "quantities and measures" using body measures, PA energy expenditure energy consumption in meals. Each proposal included description, required material, alternative, observations and supporting texts. Teachers who could not attend the training also had access to the manual and could participate in other stages of formation.

Teachers were encouraged to make the activities during the semester that were discussed during training, or create and implement similar strategies in the classroom. In general, the activities performed in the classroom included text production, videos/posters/booklets production and exposition with health issues content. The issues content in the manual could be suitable for the interests and expertise of teachers and patients (students) as well as the structural conditions of each school. A social page was created in order to monitor, assist and promote activities among teachers from the intervention schools. Finally, a meeting with the teachers of each school was made at the end of the semester to discuss the implementation of these activities.

Training and activities in Physical Education classes:

Investigators conducted a four-hour training specified to the Physical Education teachers at the beginning of school semester. Theachers were instructed to structure the predominantly active Physical Education classes, even in classes with theoretical content purposes. For example, a class focused on PA types and the relation between PA and healthy diet would be structured with a dynamic way. Investigators considered this because the active time in Physical Education classes can be a beneficial factor to total PA and adolescent health.

A supplemental manual with lesson plans and handouts was also developed and distributed to teachers. This manual was built for the program staffs and was organized by grades (7-9 grades). Materials from the Educação Física+ Project, Physical Education-specific National Curriculum Standards and health issues were used to create the manual. The manual included four units with different chapters: (i) PA and health (e.g., PA and leisure, cooperative games, PA with parents); (ii) health factors (e.g., excessive sedentary time, diabetes, hypertension, quality of life); (iii) sports (e.g., athletics, volleyball, functional training, fights); and (iv) popular games (e.g., games and dance, adventure sports). The production of posters and texts by the patient (students) with health issues content was performed as classwork or homework.

All Physical Education classes (20 classrooms with two Physical Education classes per week) during the semester were supported by a undergraduate Physical Education student. This staff collaborated in the planning of activities, material procurement organization and implementation of lessons. Additionally, one Physical Education-related event (e.g., dance festival or games competitions) were organized in order to combine Physical Education classes and school cultural events (e.g., student's week) and to encourage the active participation during school events.

Active opportunities in school environment:

These intervention strategies aimed to promote PA opportunities within the school and stimulate it in out-school time, as well as disseminate information on the importance of an active and healthy lifestyle. Supervised and unsupervised activity were considered. Some of these strategies were focus on the engagement of girls - a high-risk subgroup for inactive lifestyle.

All these strategies were implemented at the beginning of the program. Staffs, implemented these strategies in the first two weeks of semester in order to guide the execution, material access and understanding of the rules of the games. During the semester, some Physical Education classes and "Gym in School" sessions were performed using these games in order to stimulate its realization during free-time at school. Explanatory banners were exposed in schools with content on the games rules and material access. Motivational (e.g., "Let's play with the friends!") and health (e.g., "Practice PA with friends is very good for health!") messages were also included in the banners.

Health education in school community:

Some of the previous strategies had an additional focus on promoting awareness about the benefits of an active and healthy lifestyle. Principally, the materials produced in the classroom in general and Physical Education classes and the banners exposed in schools.

Additionally, pamphlets with messages on active and healthy lifestyle were distributed at intervention schools. The program team made these pamphlets and they based on other materials programs. The content was adapted to the program objectives and local reality. Teachers and professionals specialized in health education to young people made the content selection. After this, marketing experts of the Municipal Education Department executed the graphical structure of the pamphlets.

The pamphlets were delivered in the first month to a member of the school administration (coordinator or director). Guidelines were passed on the objectives of the pamphlets and as they could be distributed. In general, the pamphlets focused on the patients (students were delivered during the early times of the school day or during classes. The pamphlets focused on parents were delivered during parents/teachers meetings or in parent visits to school. Teachers were encouraged to use the pamphlets during lessons with health messages.

ELIGIBILITY:
Inclusion Criteria:

* All six full-time schools with the program called Programa Saúde na Escola in Fortaleza were eligible
* students of both sexes
* students aged 12-15 years
* students who are enrolled in 7-9 grade classes

Exclusion Criteria:

* students who are younger than 12 years-old and older than 15 years-old
* students with uncompleted data at baseline or 4-months follow-up
* students who are absence in the school days with data collection
* students who dropout the school
* students who refused to participate in data collection or intervention

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1085 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in weekly time in moderate-to-vigorous physical activity at 4 months | baseline and after 4-months of intervention
  A list of 24 types of PA will be used to measuring the weekly frequency and the daily duration of each PA that the patients perform in a typical week. Thus, the weekly PA volume and the chance in this score for each patient will be calculated.
Change from baseline in the daily time using TV/computer/video games at 4 months | baseline and after 4-months of intervention
  The daily time using TV/computer/video games of the patient will be estimated at baseline and after 4 months of intervention and the chance in this score for each patient will be calculated.

SECONDARY OUTCOMES:
Change from baseline in the healthy eating score at 4 months | baseline and after 4-months of intervention
  Healthy eating score will be estimated using three items related to healthy foods (fruit juice, fruits and vegetables) and three unhealthy (soft drinks, savory and sweets) foods in a typical week. Points from this list will be estimated at baseline and after 4 months of intervention and the chance in this score for each patient will be calculated.
Change from baseline in the body mass index at 4 months | baseline and after 4-months of intervention
  Body weight (kg) and height (m) will be used to calculate the body mass index (weight/height², kg/m²). Difference between baseline and after 4 months of intervention will be calculated.
Change from baseline in the waist circumference at 4 months | baseline and after 4-months of intervention
  Difference in the waist circumference (cm) between baseline and after 4 months of intervention will be calculated.
Change from baseline in the quality of life score at 4 months | baseline and after 4-months of intervention
  The quality of life will be measured using the World Health Organization Quality of Life instrument (poor, regular, good, great). Difference in this score between baseline and after 4 months of intervention will be calculated.
Change from baseline in the self-rated health score at 4 months | baseline and after 4-months of intervention
  The self-rated health will be measured using the World Health Organization Quality of Life instrument (poor, regular, good, great). Difference in this score between baseline and after 4 months of intervention will be calculated.
Change from baseline in the stress score at 4 months | baseline and after 4-months of intervention
  Stress will be measured using a item about stress in patients' life. Difference in this score between baseline and after 4 months of intervention will be calculated.
Change from baseline in the sleepiness score at 4 months | baseline and after 4-months of intervention
  The sleepiness (i.e., chance of dozing or sleeping) in eight patients' living situations (e.g., studying, talking, commuting to school) will be considered. Difference in this score between baseline and after 4 months of intervention will be calculated.
Change from baseline in the academic performance score at 4 months | baseline and after 4-months of intervention
  Standardized tests, academic achievement and school attendance will be evaluated in order to create an academic performance score. Difference in this score between baseline and after 4 months of intervention will be calculated.
Change from baseline in the depression scale at 4 months among obese patients | baseline and after 4-months of intervention
  Depressive symptoms will be evaluated using the scale proposed by Silveira and George at baseline and after 4 months of intervention among obese patients (World Health Organization Criteria for children and adolescents). Difference in this score between baseline and after 4 months of intervention will be calculated.
Change from baseline in the eating disorders scale at 4 months among obese patients | baseline and after 4-months of intervention
  Eating attitudes disorders will be assessed using the Eating Attitudes Test (EAT-26) at baseline and after 4 months of intervention among obese patients (World Health Organization Criteria for children and adolescents). Difference in this score between baseline and after 4 months of intervention will be calculated.
Change from baseline in the objectively-measured physical activity time at 4 months among obese patients | baseline and after 4-months of intervention
  The weekly time in physical activity will be measured objectively using the ActiGraph GT1M accelerometers in the left wrist during seven consecutive days at baseline and after 4 months of intervention among obese patients (World Health Organization Criteria for children and adolescents). Difference in this physical activity time between baseline and after 4 months of intervention will be calculated.
Change from baseline in the body image score at 4 months | baseline and after 4-months of intervention
  The self-assessment of the nine-silhouettes scale proposed by Stunkard et al. will be used to create the body image score. Difference in this score between baseline and after 4 months of intervention will be calculated.

OTHER OUTCOMES:
Change from baseline in the score of intrapersonal PA mediators at 4 months | baseline and after 4-months of intervention
  Points obtained from a list of attitude (5 items), expectations (10 items) and self-efficacy (12 items) variables will be estimated at baseline and after 4 months of intervention and the chance in this score for each patient will be calculated.
Change from baseline in the score of interpersonal PA mediators at 4 months | baseline and after 4-months of intervention
  Points obtained from a list of parental support (7 items), friends support (6 items) and teachers support (6 items) scale will be estimated at baseline and after 4 months of intervention and the chance in this score for each patient will be calculated.
Change from baseline in the score of environmental PA mediators at 4 months | baseline and after 4-months of intervention
  Points obtained from a list of perceived neighborhood environment (16 items) and school environment (7 items) scale will be estimated at baseline and after 4 months of intervention and the chance in this score for each patient will be calculated.
Change from baseline in the score of intrapersonal screen time use mediators at 4 months | baseline and after 4-months of intervention
  Points obtained from a list of attitude (3 items), expectations (12 items) and self-efficacy (11 items) variables will be estimated at baseline and after 4 months of intervention and the chance in this score for each patient will be calculated.
Change from baseline in the score of interpersonal screen time use mediators at 4 months | baseline and after 4-months of intervention
  Points obtained from a list of family and friends modelling (4 items), social support (4 items) and family norms (6 items) variables will be estimated at baseline and after 4 months of intervention and the chance in this score for each patient will be calculated.
Change from baseline in the score of environmental screen time use mediators at 4 months | baseline and after 4-months of intervention
  Points obtained from a list of family environment (8 items), school environment (4 items) and environmental characteristics (8 items) will be estimated at baseline and after 4 months of intervention and the chance in this score for each patient will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Adair S LOPES, PhD, Principal Investigator — Federal University of Santa Catarina

REFERENCES:
- [Derived] Bandeira ADS, Silva KS, Bastos JLD, Silva DAS, Lopes ADS, Barbosa Filho VC. Psychosocial mediators of screen time reduction after an intervention for students from schools in vulnerable areas: A cluster-randomized controlled trial. J Sci Med Sport. 2020 Mar;23(3):264-269. doi: 10.1016/j.jsams.2019.09.004. Epub 2019 Sep 13. PMID 31543460
- [Derived] Barbosa Filho VC, Bandeira ADS, Minatto G, Linard JG, Silva JAD, Costa RMD, Manta SW, Sa SAM, Matias TS, Silva KSD. Effect of a Multicomponent Intervention on Lifestyle Factors among Brazilian Adolescents from Low Human Development Index Areas: A Cluster-Randomized Controlled Trial. Int J Environ Res Public Health. 2019 Jan 18;16(2):267. doi: 10.3390/ijerph16020267. PMID 30669291
- [Derived] Barbosa Filho VC, da Silva KS, Mota J, Vieira NFC, Gubert FDA, Lopes ADS. "For whom was it effective?" Moderators of the effect of a school-based intervention on potential physical activity determinants among Brazilian students. Prev Med. 2017 Apr;97:80-85. doi: 10.1016/j.ypmed.2017.01.007. Epub 2017 Jan 19. PMID 28111095
- [Derived] Barbosa Filho VC, Lopes Ada S, Lima AB, de Souza EA, Gubert Fdo A, Silva KS, Vieira NF, Trompieri Filho N, de Araujo TS, de Bruin PF, Mota J; "Fortaleca sua Saude" Working Group. Rationale and methods of a cluster-randomized controlled trial to promote active and healthy lifestyles among Brazilian students: the "Fortaleca sua Saude" program. BMC Public Health. 2015 Dec 7;15:1212. doi: 10.1186/s12889-015-2543-2. PMID 26643919
- Available data/document: Study Protocol — https://bmcpublichealth.biomedcentral.com/articles/10.1186/s12889-015-2543-2 — Study design paper
- Available data/document: Individual Participant Data Set — http://www.scielo.br/scielo.php?pid=S1980-00372016000200207&script=sci_arttext — Instrument validation study
- Available data/document: Individual Participant Data Set — http://journals.humankinetics.com/doi/abs/10.1123/jpah.2016-0113 — Intervention results